CLINICAL TRIAL: NCT01534572
Title: Significance of Synbiotics on Inflammation and Proliferation of Colonic Mucosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 538/2005
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics_Lactobacillus (Experimental): Intervention (2 weeks) with a strain of Lactobacillus
  Interventions: Dietary Supplement: Lactobacillus
- Probiotics_Bifidobacterium (Experimental): Intervention (2 weeks) of daily supplementation of a probiotic strain of Bifidobacterium.
  Interventions: Dietary Supplement: Bifidobacterium

INTERVENTIONS:
Dietary Supplement: Lactobacillus — Intervention (2 weeks) with a strain of Lactobacillus
  Other Names: Lactobacillus plantarum
  Arms: Probiotics_Lactobacillus
Dietary Supplement: Bifidobacterium — Intervention (2 weeks) with a strain of Bifidobacterium
  Other Names: Bifidobacterium infantis
  Arms: Probiotics_Bifidobacterium

SUMMARY:
There is a constant exchange between the gut epithelium and lumen, including microbial interplay. The aim of this study was to investigate dietary test products on inflammatory proliferation markers in the gut, and thereby if the products had positive effects in the gut as well as in other parts of the body.

The hypothesis was that the test products would reduce the inflammatory and proliferation activity of the gut epithelium by fermentation of normal food products and by converting dietary phenolic compounds into anti-inflammatory substances.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old,
* Able to understand oral and written information,
* Informed consent

Exclusion Criteria:

* Ongoing immune suppressive treatment, incl. cortisone,
* Ongoing antibiotic treatment or antibiotic treatment ended within 4 weeks,
* History of inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reactivity of rectal mucosa | after 2 weeks intervention
  to study the reactivity of rectal mucosa after a standardized inflammatory insult before and after treatment with probiotics

SECONDARY OUTCOMES:
influence on immune system | after 2 weeks intervention
  to study the influence on systemic leukocytes and regulatory T cells

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Jeppson, MD, PhD, Study Director — Region Skåne

REFERENCES:
- [Derived] Stene C, Rome A, Palmquist I, Linninge C, Molin G, Ahrne S, Johnson LB, Jeppsson B. Administration of probiotics to healthy volunteers: effects on reactivity of intestinal mucosa and systemic leukocytes. BMC Gastroenterol. 2022 Mar 5;22(1):100. doi: 10.1186/s12876-022-02185-1. PMID 35247974